CLINICAL TRIAL: NCT05561504
Title: HelicoPTER - Bestimmung Der Lokalen Helicobacter Pylori Prävalenz Und Antibiotika Resistenzlage
Brief Title: Helicobacter Pylori Local Prevalence and Antibiotic Resistance
Acronym: HelicoPTER
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: GI 06.827
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Gastritis; Drug Resistant Bacterial Infection; Antibiotic Resistant Infection; Gastric Cancer; Microbial Colonization
MeSH Terms: conditions — Stomach Neoplasms; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, fecal samples, gastric biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical management of H. pylori infection depends essentially on two factors, prevalence and local resistance. In Germany, only limited data from rather small cohorts currently exist regarding both factors. Knowledge of the current prevalence (accounting for socioeconomic factors and age) is important for the selection of suitable detection methods, as this influences the positive and negative predictive value of the respective diagnostic methods. Current data on antibiotic resistance are essential for efficient therapy. In this clinical study, we will collect data on the frequency and severity of H. pylori infections and then, after endoscopic examination, on antibiotic resistance. Knowledge of the resistance situation is necessary for the selection of suitable therapeutic regimens. Furthermore, molecular methods for resistance detection are to be compared with conventional microbiological methods in order to be able to detect resistance more quickly. Furthermore, we aim to identify specific parameters for early detection of patients at particularly high risk of gastric cancer or with precancerous lesions due to infection. The aim is to identify carcinogenesis-relevant factors such as gastric microbiome signatures that will make it possible to identify patients who are most likely to benefit from prophylactic eradication therapy in terms of risk stratification.

DETAILED DESCRIPTION:
Infection with H. pylori occurs in childhood and usually leads to lifelong persistence of the pathogen. The prevalence of the infection depends on socioeconomic status (occupation, income, housing situation), especially during childhood, when the transmission occurs most frequently. H. pylori infections are most common in East Asia, e.g. China, with prevalence rates of around 60-80 %, and in Africa, with prevalence rates of partly over 80 %. In Europe, there is a south-north divide in infection rates with a higher prevalence in southern countries. The prevalence in Germany varies between 21% for the Hannover area and 44% for Saxony-Anhalt; the prevalence in children is significantly lower than in adults. Current data on the larger population in Germany are lacking. While antibiotics in combination with PPIs can be used to treat the infection, rising antibiotic resistance rates reduce effectiveness of eradication regimens.

We therefore initiated a multicenter observational study to assess the prevalence of H. pylori infection and antibiotic resistance rates in Germany. In Part A, volunteers are screened for H. pylori infection by serology. If the test is positive, a breath test is performed for confirmation and further visits and examinations follow for long-term observation. Positive patients undergoing endoscopy can enter Part B, in which biopsies are taken for antibiotic resistance, and establishment of a serum, stool and a tissue bank for molecular analysis including microbiome sequencing.

Part A - Primary study objectives - screening phase The primary aim of this part of the study is to collect data on the prevalence of H. pylori in an age- and gender-stratified random sample of the populations of Munich, Tübingen, Hannover, Regensburg, and Magdeburg and their respective surroundings. If the initial serologic test is negative, no further study visits are planned for these subjects. The serum samples already collected will be used as control samples for the serologic study. If the serologic test is positive, a breath test is performed for confirmation. If the confirmatory breath test is positive and the subject is evaluated by his/her primary doctor and deemed a candidate for endoscopic evaluation, then s/he is referred for participation in part B of the study.

Part B - Secondary study objectives - investigation phase

As secondary study objectives, the following should be investigated in H. pylori infected study participants:

* Establishment of a patient cohort for long-term observation (5-10 years).
* Establishment of a serum, stool and tissue bank in this cohort for subsequent testing:

  * H. pylori subtype determination for gastric cancer risk, early detection via antibody responses in serum, identification of risk factors
  * PCR or sequencing of H. pylori strains (from stomach biopsy or stool sample)
  * H. pylori isolation and antibiotic resistance testing from gastric mucosa biopsies, only to be performed as part of a clinically indicated esophago-gastro- duodenoscopy - ÖGD (for diagnosis before initiation of therapy or also after completion of therapy to monitor success or progression)
  * Correlation of microbiological findings with histopathological findings and atrophy markers.
* Determination of H. pylori associated microbiome characteristics and microbiome changes after eradication therapy

Only patients undergoing gastroscopy for clinical indications are included into Part B of the study

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* informed consent for HelicoPTER study
* informed consent for HEPY biobank

Exclusion Criteria:

* no capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: unselected group of participants
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori prevalence | 6 months
  Prevalence of H. pylori infection in a random sample of the populations of Munich, Tübingen, Hannover, Regensburg, Magdeburg and their respective surroundings
H. pylori resistance profiles | 6 months
  H. pylori isolation and antibiotic resistance testing from gastric mucosa biopsies

SECONDARY OUTCOMES:
H. pylori strain analyses | 1 year
  H. pylori subtype determination via antibody responses in serum and sequencing of H. pylori strains
subsequent medical events | 10 years
  survey-based follow up of participants at 5 and 10 years for subsequent medical conditions
risk factors for gastric cancer | 10 years
  Correlation of microbiological and serological findings with gastric histopathology and subsequent cancer diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Markus Gerhard, Prof., Principal Investigator — Technical University of Munich
Locations (1):
- Department of Medicine II, University Hospital of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available after closing of recruitment (12/2025) for a duration of 10 years
Access Criteria: data transfer request with detailed outline of scientific questions and aims